CLINICAL TRIAL: NCT06088927
Title: Long-term Outcomes of Conduction System Pacing: a National Multicenter Observational Study - NORMAND'HIS / STIMU'HIS
Acronym: STIMU'HIS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/0417/OB
Record Dates: First submitted 2023-05-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-03

CONDITIONS: Conduction System Pacing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Conduction system pacing — Conduction system pacing (His Bundle Pacing or Left Bundle Branch Area Pacing)

SUMMARY:
This prospective multicenter registry will evaluate the long-term electrical, echocardiographic, and clinical outcomes of conduction system pacing (CSP). There is currently limited data in the literature regarding the long-term results and benefits of CSP. The long-term maintenance of conduction system (His bundle or Left Bundle Branch) capture and physiological ventricular activation is an essential prerequisite for the expected benefits of this technique.

There is currently no prospective study evaluating the preservation of CSP during long-term follow-up. The design of the present study will allow reliable evaluation of CSP maintenance at 2 years follow-up. The prospective collection of electrical data (pacing thresholds, impedance, R wave sensing) during pacemaker follow-up visits will confirm thresholds stability over the long term. The incidence of atrial fibrillation episodes will also be precisely evaluated and will provide new information. Although pathophysiological studies have demonstrated less impairment of left atrial function with conduction system pacing, there is currently no data on the incidence of atrial fibrillation in patients implanted with a CSP pacemaker.

Echocardiographic data will be prospectively collected in order to analyse the evolution of left ventricular ejection fraction (LVEF) after CSP. This systematic follow-up is rarely found in CSP studies, often retrospective, with significant missing echocardiographic data. The hypothesis is that patients benefiting from CSP will not develop the deleterious effects demonstrated with conventional right ventricular pacing, such as left ventricular dilation and LVEF impairment. Inter- and intraventricular asynchrony criteria will also be systematically evaluated during follow-up echocardiography.Finally, this prospective cohort will also systematically collect clinical follow-up data (hospitalizations for heart failure and NYHA stage).

ELIGIBILITY:
Inclusion Criteria:

* Patient who had undergone conduction system pacing attempt
* Age > 18 yo
* Capacity to understand the nature of the study, legal ability and willingness to give informed consent

Exclusion Criteria:

* Patient under guardianship, trusteeship, or legal protection.
* Pregnant woman (positive urine pregnancy test) or breastfeeding or lack of proven effective contraception (according to the WHO definition) or menopausal without confirmed diagnosis (non-medically induced amenorrhea for at least 12 months before the inclusion visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients referred for conduction system pacing
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from major adverse events | 24 months
  Major adverse events are defined as follow :
  * Lead revision (including infection and pacing threshold increase)
  * Lead dislodgment
  * Loss of conduction system pacing (i.e. loss of His Bundle Pacing or Left Bundle Branch area pacing according to standard definitions)
  * Heart Failure Hospitalization
  * Upgrade to BiVentricular pacing
  * All cause mortality

SECONDARY OUTCOMES:
LVEF (%) | 24 months
AF incidence | 24 months
Heart Failure Hospitalization Incidence | 24 months
CSP Threshold during pacemaker check (Volt @ ms) | 24 months
Paced QRS width | 24 months
Interventricular dyssynchrony parameters | pre-discharged
  Aortic pre-ejection time (ms) - Pulmonary pre-ejection time (ms) (echocardiography)
Intraventricular dyssynchrony parameters | pre-discharged
  Difference between the first and last left ventricular systolic peak using 2D speckle tracking (echocardiography)

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Caen, Caen
  - CHI Elbeuf, Elbeuf
  - Groupe Hospitalier La Rochelle Ré-Aunis, La Rochelle
  - CH Le Havre, Le Havre
  - CHU Lille, Lille
  - Hôpital Saint Philibert, Lomme
  - CHU Rennes, Rennes
  - Rouen University Hospital, Rouen
  - Clinique Saint Hilaire, Rouen
  - CHU Sud Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No